CLINICAL TRIAL: NCT06886516
Title: ADAPTiON: Apixaban Dose Adjustment in Patient With Thrombocytopenia in ONcology
Brief Title: Apixaban in Thrombocytopenia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rushad Patell (Other)
Responsible Party: Sponsor-Investigator, Rushad Patell, Sponsor Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-110
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism and Thrombosis; Thrombocytopenia; Recurrent Venous Thromboembolism
Keywords: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism; Thrombocytopenia; Thromboembolism; Recurrent Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis; Thrombocytopenia; Venous Thromboembolism; Thromboembolism | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DOSE-ADJUSTED APIXABAN (Experimental): 30 enrolled participants will complete study procedures as follows:
  * Baseline visit with assessments
  * Predetermined dose of Apixiban 2x daily for 90 days
  * Off treatment visit 7 days after last study drug dose
  * Follow up visit 6 weeks after last study drug dose
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — A factor Xa inhibitor, 2.5 and 5 mg tablets, by mouth per protocol.
  Other Names: 1-(4methoxyphenyl)-7-oxo-6-[4-(2-oxopiperidin-1-yl)phenyl]-4,5,6,7-tetrahydro-1H-pyrazolo[3,4c]pyridine-3-carboxamide; C25H25N5O4

SUMMARY:
This study is being done to determine the feasibility and safety of using a novel dose adjusted apixaban for the management of participants with cancer-associated venous thromboembolism (blood clot) or and thrombocytopenia (low number of platelets in the blood). Investigators are also looking to see if participants on this treatment have fewer bleeding episodes.

The name of the study drug involved in this study is:

-Apixiban (a type of anticoagulant)

DETAILED DESCRIPTION:
This study is being done to determine the feasibility and safety of using a novel dose adjusted apixaban for the management of participants with cancer-associated venous thromboembolism (blood clot) or and thrombocytopenia (low number of platelets in the blood).

This study is a feasibility study, which is the first-time investigators are examining this drug, Apixaban, for cancer-associate VTE or thrombocytopenia. Investigators are also looking to see if participants on this treatment have fewer bleeding episodes.

The U.S. Food and Drug Administration (FDA) has approved apixaban as a treatment option for venous thromboembolism (VTE) and stroke prevention in patients with atrial fibrillation (irregular and fast heartbeat). This study is investigating apixaban taken by mouth (with adjusted doses) as a treatment for VTE in participants with active malignancies (cancer) and thrombocytopenia which has not been studied or FDA approved.

The research study procedures include screening for eligibility, in-clinic visits, and blood tests.

Participants will receive study treatment for 90 days and will be followed for 6 weeks after stopping study treatment.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Active malignancy defined as histologically confirmed diagnosis within last 6 months or received any cancer directed therapy within the last 6 months.
* Radiologically confirmed newly diagnosed symptomatic deep vein thrombosis or pulmonary embolism within 28 days of enrollment. Includes proximal lower-limb DVT or symptomatic PE. Upper extremity or catheter-associated thrombosis will be included, as will distal lower extremity DVTs.
* Platelet count < 75,000/ml (prior to platelet transfusion) within 28 days of VTE diagnosis.
* Platelet count responsive to transfusion if previously administered (defined as an average platelet increase of at least 10,000/ml over the last 3 transfusions.
* No evidence of active hemorrhage.
* No recent history of major hemorrhage (requiring transfusion, hospitalization or intervention) within the last 12 months.
* No known brain metastases.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of apixaban in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤2
* Participants must have adequate organ and marrow function as defined below:

  * Total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * Glomerular filtration rate (GFR) ≥25 mL/min/1.73/m2
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* The effects of apixaban on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of apixaban administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* Participants who have had a thrombectomy, insertion of a caval filter, or require a fibrinolytic agent.
* Participants that have index events with severe clot burden defined as bilateral proximal lower extremity deep vein thrombosis and saddle embolism or pulmonary embolism with hemodynamic compromise.
* Participants with acute myeloid leukemia or myelodysplastic syndrome or who are undergoing or have undergone allogeneic stem cell transplant.
* Participants with luminal gastrointestinal malignancy or genitourinary cancer.
* Presence of known or prior brain metastasis, given the increased risk of life-threatening intracranial hemorrhage with anticoagulant use. While screening for brain metastases is not standard of care in this population, investigators may obtain brain imaging if clinically indicated prior to initiation of anticoagulation. Imaging is not mandated in order to participate in this study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to apixaban.
* Participants receiving any medications or substances that are inhibitors or inducers of CYP3A/P-gp are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Participants on aspirin (>100 mg/day), dual antiplatelet therapy, or receiving chronic treatment with NSAIDS
* Participants with uncontrolled intercurrent illness.
* Participants at high risk of bleeding such as:

  * Unresected luminal/mucosal GI and GU cancers
  * Active gastric or duodenal cancer
  * History of major bleeding (based on ISTH criteria) in the past 12 months
  * Any prior history of Intracranial hemorrhage (microhemorrhage is not included)
  * Clinical or laboratory concern for ongoing DIC (prolonged PT/APTT or low fibrinogen)
* Severe renal disease (CKD Stage IV or higher) or liver disease (Child Pugh B/C)
* Participants with pre-planned major surgery within the study period
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because apixaban has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with apixaban, breastfeeding should be discontinued if the mother is treated with apixaban.
* Participant must be able to swallow pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Study Enrollment | Up to 5 years
  Study enrollment is defined as documentation of informed consent for participants approached.

SECONDARY OUTCOMES:
Rate of Enrolled Participants With Administration of at Least 1 Dose of Apixaban | Up to 3 months
  Feasibility is achieved if 75% of participants received at least 1 dose of apixaban.
Study Drug Adherence Rate | Up to 3 months
  Study drug adherence is defined as the proportion of participants that take over 80% of prescribed doses based on pill count. Success is defined as 75% or above.
Platelet Count Monitoring Plan Adherence Rate | Up to 3 months
  Platelet Count Monitoring Plan Adherence Rate is defined as proportion of participants that receive at least 80% of platelet counts within frequency stipulated by the study protocol. Success is defined as 75% or above.
Study Completion Rate | Up to 3 months
  Study is completed when participants finish the 90-day period or terminate due to event that qualifies as an outcome.
Major Bleeding Rate | Up to 3 months
  Major bleeding rate is defined as the proportion of participants who experience major bleeding during the study.
Clinically Relevant Non-Major Bleeding Rate | Up to 3 months
  Clinically relevant major bleeding rate is defined as the proportion of participants who experience a clinically relevant non-major bleeding event.
Recurrent Venous Thromboembolism Rate (VTE) | Up to 3 months
  Recurrent VTE rate is defined as the proportion of participants who experience recurrent VTE, including pulmonary embolism and lower extremity deep vein thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Rushad Patell, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu